CLINICAL TRIAL: NCT03600623
Title: Neoadjuvant Folfirinox or Gemcitabine-Nab Paclitaxel Followed by Stereotactic Body Radiotherapy (SBRT) for Patients With Locally Advanced Pancreatic Cancer
Brief Title: Folfirinox or Gemcitabine-Nab Paclitaxel Followed by Stereotactic Body Radiotherapy for Locally Advanced Pancreatic Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI left the institution; no further accruals
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ravi Kumar Paluri, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB160830003 (UAB 1632); NCT03641183 (obsolete NCT alias)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Locally Advanced Pancreatic Cancer; Borderline Pancreatic Inoperable Cancer; Pancreatic Cancer
Keywords: advanced pancreatic cancer; inoperable pancreatic cancer; Folfirinox; Gemcitabine-Abraxane; Gemcitabine-nab-Paclitaxel; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Leucovorin; Oxaliplatin; Irinotecan; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to one of two treatment arms: Arm 1 is Folfirinox (5FU/Leucovorin/Irinotecan/Oxaliplatin) and Arm 2 is Gemcitabine-nab-Paclitaxel (Abraxane). Either arm will be followed with SBRT for eligible patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Folfirinox + SBRT (Experimental): Folfirinox comprises the following: Fluorouracil 2,400 mg/m2 intravenously over 48 hours Days 1-3 and 15-17 every 4 weeks; Folinic acid 400 mg intravenously on Days 1 and 15 every 4 weeks; Oxaliplatin 85 mg/m2 intravenously on Days 1 and 15 every 4 weeks; and Irinotecan 180 mg/m2 intravenously on Days 1 and 15 every 4 weeks. Radiation will begin at the completion of cycle 2 if chemotherapy toxicity permits and will last over a period of 5 days.
  Interventions: Drug: Folfirinox
- Gemcitabine-nab Paclitaxel + SBRT (Experimental): Gemcitabine-nab Paclitaxel comprises the following: Gemcitabine 1000 mg/m2 on Days 1, 8, and 15 every 4 weeks; nab Paclitaxel 125 mg/m2 on Days 1, 8, and 15 every 4 weeks. Radiation will begin at the completion of cycle 2 if chemotherapy toxicity permits and will last over a period of 5 days.
  Interventions: Drug: Gemcitabine nab-Paclitaxel

INTERVENTIONS:
Drug: Folfirinox — SBRT will follow Folfirinox at the completion of Cycle 2 (if eligible).
  Other Names: Folfirinox = Fluorouracil + Folinic Acid + Oxaliplatin + Irinotecan
  Arms: Folfirinox + SBRT
Drug: Gemcitabine nab-Paclitaxel — SBRT will follow Gemcitabine nab-Paclitaxel at the completion of Cycle 2 (if eligible).
  Other Names: Paclitaxel = Abraxane
  Arms: Gemcitabine-nab Paclitaxel + SBRT

SUMMARY:
This study will implement a new treatment regimen for patients with advanced and inoperable pancreatic cancer using chemotherapy combinations of Folfirinox or gemcitabine-nab paclitaxel (abraxane) followed by a short course of high dose radiation called Stereotactic Body Radiation Therapy (SBRT). While the chemotherapy is standard of care, the strategy of adding SBRT has not been investigated. An increase in the percentage of patients who can proceed to have surgery to remove their disease is anticipated with this approach.

DETAILED DESCRIPTION:
This pilot study will evaluate safety and tolerability of neoadjuvant chemotherapy followed by SBRT. Patients with locally advanced pancreatic cancer (LAPC) and borderline pancreatic inoperable cancer will be assigned to one of two treatment arms based upon performance status and physician's discretion. The two treatment arms are: Folfirinox or gemcitabine-nab paclitaxel (abraxane). There are no study drugs as all treatments are based on standard clinical pathways.

After two cycles of treatment patients will be restaged with CT scans or imaging. If the tumor remains resectable, borderline, or unresectable without progression of disease, then the patient will proceed to SBRT.

Follow-up visits will continue every three months for up to one year or until progression of disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the pancreas. Patients with mixed tumor with predominant adenocarcinoma pathology can be enrolled.
* Subjects will be staged according to the 2010 American Joint Committee on Cancer (AJCC) staging system with pathologic stage T1-4, being eligible; and have a primary tumor of the pancreas (either pancreatic head, neck, uncinate process, or body/tail)
* The tumor must be deemed as being borderline/unresectable. Final CT confirmation of surgical staging/ eligibility will be at the discretion of the pancreatic surgeon of the patient.
* Disease must be confined to loco-regional site as confirmed by CT imaging and/or diagnostic staging laparoscopy to avoid occult peritoneal deposits. Diagnostic laparoscopy will be performed only if absolutely required
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) on imaging studies CT
* Karnofsky performance status greater than or equal to 70 or Eastern Cooperative Oncology Group (ECOG) performance of 0-2.
* Age >18
* Estimated life expectance >12 weeks
* If female patient is of child bearing potential, she must have a negative serum pregnancy test (βhCG) documented up to 72 hrs prior to administration of first study drug
* Patient has screening blood work performed which includes the following (should be drawn ≤14 days prior to enrollment)
* Absolute neutrophil count (ANC) >1.5 x 109/L
* Platelet count ≥100,000/mm3
* Hemoglobin (Hgb) ≥ 9g/dL
* Aspartate aminotransferase (AST), Alanine Aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN) Total Bilirubin ≤1.5 ULN
* Serum Cr within normal limits (WNL)
* Prothrombin Time and International Normalized Ratio (PT/INR) and Partial Thromboplastin Time (PTT) within normal limits (±15%).
* Disease must be encompassed in a reasonable SBRT "portal" as defined by the treating radiation oncologist

Exclusion Criteria:

* Ineligible Histology including non-adenocarcinomas, adenosquamous carcinoma, islet cell carcinomas, cystadenomas, cystadenocarcinomas, carcinoid tumors, duodenal carcinomas, distal bile duct and ampullary carcinomas
* Patients must not have received prior pancreatic surgery, radiation therapy, chemotherapy or any investigational therapy for pancreatic cancer.
* Patients with tumors extending or invading duodenum or gastric are not eligible.
* Evidence of distant metastasis on upright chest x-ray, CT or other staging studies
* Subjects with recurrent disease are not eligible
* Prior radiation therapy to the upper abdomen or liver at the discretion of the treating radiation oncologist could impair delivery of the prescribed radiation treatment
* Patients with scleroderma, ulcerative colitis or other systemic conditions deemed risky for radiation treatment. Therefore, will be excluded.
* Prior chemotherapy
* Subjects in their reproductive age who are breast feeding or have a positive pregnancy test
* Any co-morbid condition such as but not limited to congestive heart failure, cardiac arrhythmia or psychiatric illness of sufficient severity to limit full compliance with the protocol per assessment by the individual treating physician
* Concurrent active infection
* No prior malignancy allowed except cervical cancer in situ, adequately treated basal cell or squamous cell carcinoma of skin or treated low risk prostate cancer
* Patient with known historical or active infection with HIV, Hepatitis B or Hepatitis C
* Patient who has undergone recent major surgery, other than diagnostic surgical procedure within 4 weeks prior to enrollment.
* Patient who has a history of allergy or hypersensitivity to any of the study drugs.
* Patients with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, interstitial pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies
* Patients with greater than grade 2 peripheral neuropathy at the time of enrollment are not eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Baseline up to two years
  Initial dose of drug until 4 weeks following completion of therapy which may or may not include SBRT and follow-up. Adverse event reporting will be graded following the National Cancer Institute of Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.

SECONDARY OUTCOMES:
Progression-free survival | Baseline up to two years
  Progression-free survival is the duration of time from study entry to time of disease progression or death, whichever comes first.
Overall survival | Baseline to two years
  Overall survival is the duration of time from study entry to time of death or the date of last contact.
Rate of preoperative chemotherapy + radiotherapy completion | Baseline to two years
  The rate will be determined from the measurement of lesions (maximum of 2 per organ with no more than 5 lesions total) from CT scans and magnetic resonance imaging within the study time frame.
Proportion of participants undergoing surgery after preoperative chemoradiation therapy | Baseline to two years
  Comparison of participants who underwent surgery versus those that did not following preoperative chemoradiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ravi K Paluri, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No